CLINICAL TRIAL: NCT02856542
Title: Real-life Evaluation of an Applicator, as a New Mode of Administration of Daivobet® Gel, on Adherence to Treatment and SAtisfaction of Patients With PSOriasis
Brief Title: Real-life Evaluation of the Daivobet® Gel Applicator
Acronym: ASAP PSO
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-DAIVOBETGEL-1284
Record Dates: First submitted 2016-07-11; First posted 2016-08-05 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis vulgaris, scalp, topical, applicator, device
MeSH Terms: interventions — calcipotriene

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: calcipotriol/betamethasone dipropionate gel in Applicator — Topical treatment of scalp using applicator device. The study as such is non-interventional as the intervention has been decided prior to and independently from the inclusion of the patient in the cohort to be observed.
  Other Names: Daivobet® gel Applicator

SUMMARY:
This study aims to describe the patient population being treated and evaluate their treatment adherence and treatment outcomes during treatment of scalp psoriasis with Daivobet® gel Applicator for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Dermatologist or general practitioner has decided to initiate treatment with Daivobet® gel Applicator

Exclusion Criteria:

* Indication not within the approved labelling in France
* Contraindication for treatment with calcipotriol or betamethasone dipropionate
* Informed consent to participate in the study has not been obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with psoriasis vulgaris affecting the scalp who are prescribed scalp treatment with Daivobet® gel Applicator.
  Representativeness is ensured through random sampling of investigators to be invited to participate from a country wide list of dermatologists and general practitioners, with adjustment for regional distribution. Investigators include their first three patients meeting the study criteria.
Sampling Method: Probability Sample
Enrollment: 1560 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Morisky Medication Adherence Scale-8 | 2 weeks
  Degree of adherence to prescribed treatment
Morisky Medication Adherence Scale-8 | 4 weeks
  Degree of adherence to prescribed treatment

SECONDARY OUTCOMES:
Patient opinion on Applicator usability | 4 weeks
  5-point Likert scale
Patient overall satisfaction | 4 weeks
  4 point Likert scale
Patient Global Impression of Improvement | 2 weeks
  7 point Likert scale
Patient Global Impression of Improvement | 4 weeks
  7 point Likert scale
Investigator's opinion on the properties of the Applicator | Baseline
  5 point rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde Kemula, MD, Principal Investigator — Cabinet de Dermatologie, Dr. Mathilde Kemula; Frederic Bonnier, MD, Principal Investigator — General Practice, 356 Rue de Charles de Gaulle, 91400 Orsay; Nathalie Quiles, MD, Principal Investigator — Hôpital Saint Joseph, 26 Boulevard de Louvain, Marseille
Locations (1):
- Cabinet de Dermatologie, Dr. Mathilde Kemula, Charenton-le-Pont, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morisky DE, Green LW, Levine DM. Concurrent and predictive validity of a self-reported measure of medication adherence. Med Care. 1986 Jan;24(1):67-74. doi: 10.1097/00005650-198601000-00007. PMID 3945130